CLINICAL TRIAL: NCT01767181
Title: Effects of Timed Intensive Light Therapy or Timed Physical Exercise on Markers of Central and Peripheral Circadian Rhythm and on Cardiometabolic Function in Night Shift Workers
Brief Title: Light and Exercise in Night-shift Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EuRhythDia-1
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Healthy Night Shift Workers
Keywords: Light therapy; physical exercise; night shift workers; genetic markers; PBMCs
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (No Intervention): Control group without intervention
- B (Experimental): Intensive light therapy during the first half of the night shift
  Interventions: Other: Intensive light therapy
- C (Experimental): Exercise before the beginning of the night shift
  Interventions: Other: Exercise
- D (Experimental): Exercise after the end of the night shift
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Intensive light therapy — Light therapy will be applied by a Lumie Brazil fluorescent tube light box (10.000 lux) during the night shifts for 12 consecutive weeks
  Arms: B
Other: Exercise — Physical exercise will be performed in a supervised environment on the days of the night shifts, either before the start of the shift (defined as a time period beginning no earlier than 2 hours before the start of the shift) or after the end of the night shift (defined as a time period ending no longer than 2 hours after the end of the night shift)
  Arms: C; D

SUMMARY:
EuRhythDia is a multicenter, controlled and randomized study. The aim of the study is to investigate the effects of 12 weeks of randomized timed light therapy or timed physical exercise as a chronotherapeutic lifestyle intervention on markers of central and peripheral circadian rhythms and cardiometabolic function in healthy night shift workers.

DETAILED DESCRIPTION:
Lifestyle interventions have been recognized as important means to prevent and treat cardiometabolic disease. However, compliance of the European population to general recommendations of exercise and weight loss is unsatisfactory. There have been no studies that have attempted to convert the exciting new experimental data on the circadian clock, lifestyle, and cardiometabolic risk into diagnostic tools or novel therapeutic approaches via structured multidisciplinary efforts. One of the aims of the EuRhytDia study is to study novel applications of established lifestyle interventions by co-ordinating the timing of interventions with circadian rhythmicity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects above the age of 18
* Night shift workers on regular night shifts with at least 3 nights in a row per month during the study period
* Subjects must have been on night shifts for at least 4 weeks before inclusion into the study
* Signed written informed consent

Exclusion Criteria:

* Regular use of drugs (prescription or non-prescription, exception: contraceptives) or dietary supplements within 4 weeks before inclusion of the study
* Pregnancy or breast feeding
* Any severe somatic or psychic disease (malignant or non-malignant
* Any known ophthalmological condition that prevents the exposure to bright light (e.g. cataract, glaucoma, retinopathy, macular degeneration, acute eye infections, lesions of the cornea)
* Any skin condition or use of drugs associated with increased photosensitivity;
* Any kind of disability that would prevent the subjects from participation in exercise training sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2013-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Efficacy | 12 weeks
  The difference of the expression pattern of the CLOCK gene in peripheral blood mononuclear cells (PBMCs) after 12 weeks between intervention and control group

SECONDARY OUTCOMES:
Efficacy | 12 weeks
  The changes in body weight, BMI, abdominal circumference from baseline to 12 weeks of intervention
Efficacy | 12 weeks
  The differences in the circadian expression pattern of genes involved in circadian rhythm (e.g., Cryptochrome 1, Bmal 1, RORα, Rev-erbα, Period 1, Period 3, Timeless, Adam 17, PPAR-α, PPAR-γ, Klotho, DDAH-1, DDAH-2, AGXT 2, AGAT, VDR, TIMP 3) in peripheral blood mononuclear cells (PBMCs) after 12 weeks between intervention and control group
Efficacy | 12 weeks
  The differences in the expression of genes involved in circadian rhythm (e.g. Cryptochrome 1, Clock, Bmal 1, RORα, Rev-erbα, Period 1, Period 3, Timeless, Adam 17, PPAR-α, PPAR-γ, Klotho, DDAH-1, DDAH-2, AGXT 2, AGAT, VDR, TIMP 3) in adipose tissue and muscle tissue, between baseline and 12 weeks of intervention (restricted to participants who consent to this part of the study
Efficacy | 12 weeks
  The reversibility of the differences in the expression profiles of genes involved in circadian rhythm in peripheral blood mononuclear cells (PBMCs) 12 weeks after the end of the intervention period (=week 24 of the study)
Efficacy | 12 weeks
  The differences in epigenetic profiles of genes involved in circadian rhythm between baseline and 12 weeks of intervention
Efficacy | 12 weeks
  The reversibility of the differences in the biochemical markers and indices of cardiometabolic function (e.g. fasting glucose, fasting insulin, HOMA, OGTT, QUICKI index, Stumvoll-ISI index, HbA1c, ADMA, SDMA, fibrinogen, PAI-1, triglycerides, total cholesterol, LDL-cholesterol, HDL-cholesterol, C-reactive protein, C3, systolic and diastolic blood pressure, endothelial function, IMT) 12 weeks after the end of the intervention period (=week 24 of the study)
Efficacy | 12 weeks
  The differences in metabolomic profiling between baseline, 12 weeks of intervention, and after 12 weeks of wash-out (Plasma samples will be collected for metabolomic analysis at these time points)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Böger, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No